CLINICAL TRIAL: NCT03570918
Title: A Phase 1 Study to Evaluate the Safety, Immunologic and Virologic Responses of MGD014 Therapy in HIV-Infected Individuals on Suppressive Antiretroviral Therapy
Brief Title: MGD014 in HIV-Infected Individuals on Suppressive Antiretroviral Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MacroGenics (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGD014-01; 272201500032C-2-0-1 (NIH)
Record Dates: First submitted 2018-06-18; First posted 2018-06-27 (Actual); Results first posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: HIV-1-infection
Keywords: HIV, Latent HIV-1 infection, HIV therapy, antibody-based therapy

STUDY DESIGN:
Intervention Model Description: Open-label dose-escalation study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- MGD014 0.1 micrograms/kilogram (mcg/kg) (Experimental): a single 2-hour infusion
  Interventions: Biological: MGD014
- MGD014 0.3 mcg/kg (Experimental): a single 2-hour infusion
  Interventions: Biological: MGD014
- MGD014 1.0 mcg/kg (Experimental): a single 2-hour infusion
  Interventions: Biological: MGD014
- MGD014 3.0 mcg/kg (Experimental): a single 2-hour infusion
  Interventions: Biological: MGD014
- MGD014 10.0 mcg/kg (Experimental): a single 2-hour infusion
  Interventions: Biological: MGD014
- MGD014 30.0 mcg/kg (Experimental): a single 2-hour infusion
  Interventions: Biological: MGD014
- MGD014 100.0 mcg/kg (Experimental): a single 2-hour infusion
  Interventions: Biological: MGD014
- MGD014 300.0 mcg/kg (Experimental): a single 2-hour infusion
  Interventions: Biological: MGD014
- MGD014 300.0 mcg/kg multiple doses (Experimental): 2-hour infusion every 2 weeks for 3 infusions
  Interventions: Biological: MGD014

INTERVENTIONS:
Biological: MGD014 — HIV-1 x CD3 bispecific DART molecule

SUMMARY:
This is a Phase 1, open-label single-center study to determine the safety of MGD014 in participants with human immunodeficiency virus (HIV) infection on stable suppressive antiretroviral therapy (ART).

DETAILED DESCRIPTION:
Eligible participants will be maintained on ART and receive either one infusion (Part 1) or multiple infusions of MGD014 (Part 2). Part 1 is a single ascending dose study with a 1+3 design for the first 2 dose cohorts, and a 3+3 design with staggered accrual for the 6 higher dose cohorts, with an aim of determining the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of ascending doses up to either the Optimal Biologic Dose (OBD) or the maximum administered dose (MAD).

Part 2 is a multi-dose expansion cohort with MGD014 administered at the OBD, as determined in Part 1. In Part 2, additional assessments on the effects of MGD014 on HIV latent infection parameters will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness of participant to provide written informed consent.
* HIV-1 infection, documented by any FDA-approved rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral load.
* On a potent, stable, continuous ART regimen for ≥ 24 months prior to Screening.
* Plasma HIV-1 RNA < 50 copies/mL at two time points in the previous 12 months prior to screening (one time point can be screening) and never ≥ 50 copies/mL on 2 consecutive time points in the last 24 months.
* Adequate organ function based on acceptable laboratory parameters.

Exclusion Criteria:

* Women of childbearing potential defined as any female who has experienced menarche and who has not undergone successful surgical sterilization or menopause.
* History or other evidence of severe illness, immunodeficiency other than HIV, or any other condition that would make the potential participant unsuitable for study.
* History or other evidence of any condition or process for which signs or symptoms could be confused with reactions to MGD014.
* History of any HIV immunotherapy or HIV vaccine except for MGD014 within 12 months prior to screening.
* History of clinically significant cardiovascular disease, severe allergic reactions, malignancy (except non-melanoma skin cancer) within 5 years, seizure disorder within 2 years, organ/tissue transplant, autoimmune disease, unstable asthma, bleeding disorder.
* Evidence of active viral, or antifungal treatment within 7 days prior to the initiation of study drug
* Active, asymptomatic, or suspected COVID-19/SARS-CoV-2 infection.
* Active, untreated syphilis.
* Use of blood products, cytokine therapy, growth-stimulating factors, cytotoxic chemotherapy or investigational therapy within 90 days.
* Current use of the antivirals maraviroc and/or enfuvirtide.
* Any vaccination with exception of flu vaccine within 30 days of screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — MacroGenics
Locations (1):
- University of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three participants who were treated in Period 1 (single dose) in the 10, 100, or 300 mcg/kg dose cohorts were also treated in Period 2 (multiple dose) in the 300 mcg/kg dose cohort.
Groups:
- MGD014 300 mcg/kg Multiple Doses: 3 infusions given every 2 weeks over 4 weeks.
Period: Period 1
Arm/Group | MGD014 0.1 Micrograms/Kilogram (mcg/kg) | MGD014 0.3 mcg/kg | MGD014 1.0 mcg/kg | MGD014 3.0 mcg/kg | MGD014 10.0 mcg/kg | MGD014 30.0 mcg/kg | MGD014 100.0 mcg/kg | MGD014 300.0 mcg/kg | MGD014 300 mcg/kg Multiple Doses
Started | 1 | 1 | 4 | 3 | 3 | 3 | 3 | 3 | 0
Completed | 1 | 1 | 4 | 3 | 3 | 3 | 3 | 3 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | MGD014 0.1 Micrograms/Kilogram (mcg/kg) | MGD014 0.3 mcg/kg | MGD014 1.0 mcg/kg | MGD014 3.0 mcg/kg | MGD014 10.0 mcg/kg | MGD014 30.0 mcg/kg | MGD014 100.0 mcg/kg | MGD014 300.0 mcg/kg | MGD014 300 mcg/kg Multiple Doses
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The 3 participants treated with multiple doses of MGD014 were also treated with single doses of MGD014 at 10, 100 and 300 mg, respectively.
Groups:
- MGD014 0.1 mcg/kg; MGD014 0.3 mcg/kg; MGD014 1.0 mcg/kg; MGD014 3.0 mcg/kg; MGD014 10.0 mcg/kg; MGD014 30 mcg/kg; MGD014 100 mcg/kg; MGD014 300 mcg/kg: Single infusion of MGD014
- Total: Total of all reporting groups
Arm/Group | MGD014 0.1 mcg/kg | MGD014 0.3 mcg/kg | MGD014 1.0 mcg/kg | MGD014 3.0 mcg/kg | MGD014 10.0 mcg/kg | MGD014 30 mcg/kg | MGD014 100 mcg/kg | MGD014 300 mcg/kg | Total
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 3 | 3 | 3 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The 3 participants treated with multiple doses of MGD014 were also treated with single doses of MGD014 at 10, 100 and 300 mg, respectively
  years
    Period 1: Single Dose | 40.0 (NA) — not applicable for a single participant | 53.0 (NA) — not applicable for a single participant | 49.8 (9.18) | 37.9 (5.51) | 56.7 (7.09) | 41.0 (10.82) | 33.7 (5.86) | 42.3 (17.10) | 44.4 (11.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Single dose: Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Single dose: Male | 1 | 1 | 4 | 3 | 3 | 3 | 3 | 3 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 1 | 1 | 3 | 3 | 2 | 3 | 3 | 3 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 7
  White | 0 | 1 | 3 | 2 | 2 | 2 | 2 | 1 | 13
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 4 | 3 | 3 | 3 | 3 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emerging Adverse Events
Description: Safety is based on evaluation of adverse events (AEs) and serious adverse events (SAEs) from the time of study drug administration through the End of Study visit.
Time Frame: up to 77 days
Measure: Count of Participants; unit: Participants
Arm/Group | MGD014 0.1 Micrograms/Kilogram (mcg/kg) | MGD014 0.3 mcg/kg | MGD014 1.0 mcg/kg | MGD014 3.0 mcg/kg | MGD014 10.0 mcg/kg | MGD014 30.0 mcg/kg | MGD014 100.0 mcg/kg | MGD014 300.0 mcg/kg | MGD014 300.0 mcg/kg Multiple Doses
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 3 | 3 | 3 | 3
Participants | 1 | 1 | 4 | 3 | 2 | 2 | 2 | 3 | 2

2. Secondary Outcome: AUC Inf: Area Under the Plasma Concentration Versus Time Curve From Time 0 to Infinity of MGD014
Description: AUCinf, area under the concentration-time curve from the time of dose extrapolated to time infinity and reflects total drug exposure
Time Frame: Study Day 0 to 42
Measure: Mean (95% Confidence Interval); unit: mcg/L*hr
Groups:
- MGD014 0.1 mcg/kg; MGD014 0.3 mcg/kg; MGD014 1.0 mcg/kg; MGD014 3.0 mcg/kg; MGD014 10.0 mcg/kg; MGD014 30.0 mcg/kg; MGD014 100.0 mcg/kg: a single IV infusion of MGD014
- MGD014 300.0 mcg/kg: a single or multiple IV infusions of MGD014
Arm/Group | MGD014 0.1 mcg/kg | MGD014 0.3 mcg/kg | MGD014 1.0 mcg/kg | MGD014 3.0 mcg/kg | MGD014 10.0 mcg/kg | MGD014 30.0 mcg/kg | MGD014 100.0 mcg/kg | MGD014 300.0 mcg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 3 | 3 | 6
mcg/L*hr | 134 [NA to NA] — not calculable for single participant | 313 [NA to NA] — not calculable for single participant | 2610 [1230 to 3990] | 6360 [5420 to 7300] | 22300 [20600 to 23900] | 50900 [43600 to 58200] | 170000 [129000 to 210000] | 497000 [445000 to 549000]

3. Secondary Outcome: Cmax: Maximum Plasma Concentration
Description: Cmax is the maximum (or peak) serum concentration of a drug in the body after the drug has been administered
Time Frame: Study Day 0
Measure: Mean (95% Confidence Interval); unit: mcg/L
Arm/Group | MGD014 0.1 mcg/kg | MGD014 0.3 mcg/kg | MGD014 1.0 mcg/kg | MGD014 3.0 mcg/kg | MGD014 10.0 mcg/kg | MGD014 30.0 mcg/kg | MGD014 100.0 mcg/kg | MGD014 300.0 mcg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 3 | 3 | 6
mcg/L | 2.9 [NA to NA] — Not calculable for 1 participant | 5.8 [NA to NA] — Not calculable for 1 participant | 24.5 [13.7 to 35.3] | 67.7 [50.3 to 85.1] | 181 [161 to 200] | 469 [390 to 548] | 1640 [1130 to 2160] | 5288.4 [4590 to 5870]

4. Secondary Outcome: Tmax: Time to Maximum Concentration
Description: Tmax is the time it takes a drug to reach the maximum concentration
Time Frame: Study Day 0
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | MGD014 0.1 mcg/kg | MGD014 0.3 mcg/kg | MGD014 1.0 mcg/kg | MGD014 3.0 mcg/kg | MGD014 10.0 mcg/kg | MGD014 30.0 mcg/kg | MGD014 100.0 mcg/kg | MGD014 300.0 mcg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 3 | 3 | 6
hours | 3.0 [NA to NA] — not calculable for one participant | 1.9 [NA to NA] — not calculable for one participant | 2.4 [1.6 to 3.1] | 2.0 [1.9 to 2.0] | 2.7 [1.9 to 3.4] | 1.9 [1.9 to 2.0] | 2.6 [1.9 to 3.4] | 2.5 [2.0 to 2.9]

5. Secondary Outcome: Ctrough: Trough Level Concentration
Description: a trough level or trough concentration (Ctrough) is the concentration reached by a drug immediately before the next dose is administered,
Time Frame: Study Day 14
Population: Mean trough concentration for the 300 mcg/kg dose is from the first MGD014 infusion (taken at Day 14) for participants (n=3) in Part 2 only. Trough concentration is not applicable for single-dose cohorts.
Measure: Mean (95% Confidence Interval); unit: mcg/L
Groups:
- MGD014 300.0 mcg/kg: multiple IV infusions of MGD014
Arm/Group | MGD014 0.1 mcg/kg | MGD014 0.3 mcg/kg | MGD014 1.0 mcg/kg | MGD014 3.0 mcg/kg | MGD014 10.0 mcg/kg | MGD014 30.0 mcg/kg | MGD014 100.0 mcg/kg | MGD014 300.0 mcg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
mcg/L |  |  |  |  |  |  |  | 320 [252 to 338]

6. Secondary Outcome: Clearance
Description: Total body clearance of the drug from plasma of MGD014
Time Frame: Study Day 0 to 42
Measure: Mean (95% Confidence Interval); unit: L/hr
Arm/Group | MGD014 0.1 mcg/kg | MGD014 0.3 mcg/kg | MGD014 1.0 mcg/kg | MGD014 3.0 mcg/kg | MGD014 10.0 mcg/kg | MGD014 30.0 mcg/kg | MGD014 100.0 mcg/kg | MGD014 300.0 mcg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 3 | 3 | 6
L/hr | 0.04 [NA to NA] — not calculable for one participant | 0.07 [NA to NA] — not calculable for one participant | 0.03 [0.02 to 0.04] | 0.05 [0.04 to 0.05] | 0.04 [0.04 to 0.05] | 0.04 [0.04 to 0.05] | 0.05 [0.04 to 0.06] | 0.05 [0.05 to 0.06]

7. Secondary Outcome: Vz: Terminal Phase Volume of Distribution of MGD014
Description: The ratio of the total quantity of drug in the body to drug plasma concentration during the elimination
Time Frame: Study Day 1, 2, 7, 14, 21, 28, and 42 (single infusion) and Study Day 1, 3, 14, 28, 42, and 77 (multiple infusions)
Measure: Mean (95% Confidence Interval); unit: liters
Arm/Group | MGD014 0.1 mcg/kg | MGD014 0.3 mcg/kg | MGD014 1.0 mcg/kg | MGD014 3.0 mcg/kg | MGD014 10.0 mcg/kg | MGD014 30.0 mcg/kg | MGD014 100.0 mcg/kg | MGD014 300.0 mcg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 3 | 3 | 6
liters | 2.1 [NA to NA] — not calculable for one participant | 4.1 [NA to NA] — not calculable for one participant. | 8.7 [6.2 to 11.2] | 19.7 [14.2 to 25.2] | 17.5 [16.9 to 18.2] | 17.4 [15.4 to 19.3] | 21.6 [16.9 to 26.2] | 15.8 [9.1 to 22.5]

8. Secondary Outcome: Terminal Half Life of MGD014
Description: The half-life is the amount of time required for 50% of the drug to be removed from the body
Time Frame: Study Day 0 to Study Day 42
Population: Average terminal half-life did not include participants in Part 2 (n=3) due to a shortened PK schedule that did not support estimation of half-life
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | MGD014 0.1 mcg/kg | MGD014 0.3 mcg/kg | MGD014 1.0 mcg/kg | MGD014 3.0 mcg/kg | MGD014 10.0 mcg/kg | MGD014 30.0 mcg/kg | MGD014 100.0 mcg/kg | MGD014 300.0 mcg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 3 | 3 | 6
hours | 32.0 [NA to NA] — not calculable for one participant | 38.6 [NA to NA] — not calculable for one participant | 244 [136 to 351] | 300 [227 to 373] | 295 [266 to 323] | 282 [276 to 288] | 285 [269 to 300] | 295 [289 to 305]

9. Secondary Outcome: Number of Participants That Developed Antidrug Antibodies to MGD014
Description: Number of participants with antidrug antibodies to MGD014
Time Frame: Study Day 1, 14, 28 and 42 (single infusion) and Study Day 1, 14, 28 and 77 (multiple infusions)
Measure: Count of Participants; unit: Participants
Arm/Group | MGD014 0.1 mcg/kg | MGD014 0.3 mcg/kg | MGD014 1.0 mcg/kg | MGD014 3.0 mcg/kg | MGD014 10.0 mcg/kg | MGD014 30.0 mcg/kg | MGD014 100.0 mcg/kg | MGD014 300.0 mcg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 3 | 3 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

10. Secondary Outcome: Number of Participants With Increased Cytokine Levels
Description: Number of participants with increased cytokine levels from baseline after MGD014 administration. This safety measure compares serum cytokine levels obtained prior to dosing with levels obtained after dosing. Increased cytokines can be a measure of T-cell activation in response to MGD014 binding. Cytokines analyzed included interferon-gamma, tumor necrosis factor-alpha, interleukin (IL)2, IL-5, IL-6, and IL-10.
Time Frame: Study Day 1, 2 and 7 (single infusion) and Study Day 1, 3, 14 and 28 (multiple infusions)
Measure: Count of Participants; unit: Participants
Arm/Group | MGD014 0.1 mcg/kg | MGD014 0.3 mcg/kg | MGD014 1.0 mcg/kg | MGD014 3.0 mcg/kg | MGD014 10.0 mcg/kg | MGD014 30.0 mcg/kg | MGD014 100.0 mcg/kg | MGD014 300.0 mcg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 3 | 3 | 6
Participants | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 19 weeks
Groups:
- Multiple Dose MGD014 300 mcg/kg: Infusion every 2 weeks for 3 infusions.
Arm/Group | MGD014 0.1 mcg/kg | MGD014 0.3 mcg/kg | MGD014 1.0 mcg/kg | MGD014 3.0 mcg/kg | MGD014 10.0 mcg/kg | MGD014 30 mcg/kg | MGD014 100 mcg/kg | MGD014 300 mcg/kg | Multiple Dose MGD014 300 mcg/kg
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/4 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/4 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 4/4 | 3/3 | 2/3 | 2/3 | 2/3 | 3/3 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MGD014 0.1 mcg/kg (N=1) | MGD014 0.3 mcg/kg (N=1) | MGD014 1.0 mcg/kg (N=4) | MGD014 3.0 mcg/kg (N=3) | MGD014 10.0 mcg/kg (N=3) | MGD014 30 mcg/kg (N=3) | MGD014 100 mcg/kg (N=3) | MGD014 300 mcg/kg (N=3) | Multiple Dose MGD014 300 mcg/kg (N=3)
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — swollen lymph nodes
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — earwax impaction
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Application site erythema (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 — Application site redness
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Vessel puncture site pain (General disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Feeling hot (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vessel puncture site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — Insect bite
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — lab measurement of kidney function decreased
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 — Joint pain
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — muscle pain
Headache (Nervous system disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Emotional distress (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/18/NCT03570918/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/18/NCT03570918/SAP_001.pdf